CLINICAL TRIAL: NCT00350753
Title: A Phase II Study of Erlotinib and Bevacizumab in Patients With Advanced Upper Gastrointestinal Carcinomas, Refractory or Intolerable to Standard Systemic Therapy
Brief Title: Avastin and Tarceva for Upper Gastrointestinal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Ulrik Lassen, Rigshospitalet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB-UGI-01; 2006-001308-35
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Cholangiocarcinoma; Gallbladder Cancer
Keywords: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

ARMS (1):
- Erlotinib and bevacizumab (Experimental)
  Interventions: Drug: Erlotinib and bevacizumab

INTERVENTIONS:
Drug: Erlotinib and bevacizumab — Erlotonib 150 mg daily bevacizumab 10 mg/kg every 14 days

SUMMARY:
Erlotinib and bevacizumab have shown activity individually, as single drugs, or in combination with chemotherapy in upper gastro-intestinal cancers, including esophageal and gastro-esophageal adenocarcinomas, gastric cancer and pancreatic cancer. Biomarkers indicating an important role of EGF and VEGF have been found in these tumors, and in cholangiocarcinomas as well. There is promise that combined treatment with erlotinib and bevacizumab is active and tolerable in a broad range of upper gastro-intestinal cancers, justifying an experimental phase II-study of patients with these diagnoses, refractory or intolerant to standard systemic therapy.

DETAILED DESCRIPTION:
Primary Objective

* To determine the median time to progression (TTP) and response rate (RR) of the combination of erlotinib and bevacizumab in patients with advanced upper gastro-intestinal carcinomas, refractory or intolerant to standard systemic therapy.

Secondary Objective

* To determine safety, tolerability and toxicity.
* To determine median and overall survival (OS).
* To correlate efficacy of treatment with the expression of tumor markers obtained in serum (EFGR, bFGF, p-VEGF-A, and sVEGF-R2), in paraffin embedded tumor tissue (micro vessel density (MVD), and expression of VEGFR and EGFR, after immunostaining), and in fresh frozen tumor biopsies (micro array-based analyses of patterns of gene expression).

Treatment:

Bevacizumab (AvastinÒ) will be given intravenously at 10 mg/kg every other week.

Erlotinib is given as an orally daily dose and most be taken at least one hour before or two hours after ingestion of food.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically verified carcinoma of the gall bladder or bile ducts.
* PS 0-1 (ECOG scale)
* Age > 18 years
* Life expectancy > 3 months
* Sufficient organ function, defined as:

  * Platelets > 100 x 109/liter
  * Leukocytes > 3,0 x 109/liter
  * ACN > 1,5 x 109/liter
  * ASAT and/or ALAT < 3 x upper normal limit
  * Bilirubin < 1,5 x upper normal limit
  * EDTA clearance > 45 ml/min
  * APTT and INR < normal limit
* Fertile females must use oral contraceptive, IUD (intrauterine device) or preservatives. Fertile males must use preservatives.

Exclusion Criteria:

* Radiotherapy or chemotherapy within the last 4 weeks
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Any prior EGFR- or VEGFR-based therapy
* Any condition (medical, social, psychological), which would prevent adequate information and follow-up
* Tumor located close to major blood vessels and judged to possess a high risk of serious bleeding
* Any other active malignancy, except basal or squamous cell carcinoma of the skin, or carcinoma in situ
* Any significant cardiac disease (New York Heart Association Class II or greater), significant arrythmia, congestive heart failure, acute myocardial infarction within 6 months or unstable angina pectoris
* Clinically significant peripheral vascular disease
* Evidence of coagulopathy
* Use of ASA, NSAIDs or clopidogrel
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to treatment, anticipation of need for major surgical procedure during the curse of the study

  o Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to treatment
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 month prior to treatment
* Any ongoing infection, uncontrolled diabetes mellitus, serious non-healing wound or ulcer
* Pregnancy or breast feeding
* Ongoing therapeutic anti-coagulation
* Hypertension with blood pressure > 150/100 mmHg

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Objective response by RECIST criteria | From time of treatment start to response evaluation
Time to progression | 1 year

SECONDARY OUTCOMES:
Toxicity evaluated by NCI-CTCae version 3.0 | 1 year
Survival | 1 year
Biomarkers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD., PH.D., Principal Investigator — Rigshospitalet, Dept. of Oncology
Locations (3):
- Denmark (3):
  - Århus Sygehus, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense